CLINICAL TRIAL: NCT04457609
Title: Application of Umbilical Cord Mesenchymal Stem Cells as Adjuvant Therapy for Critically-Ill COVID-19 Patients
Brief Title: Administration of Allogenic UC-MSCs as Adjuvant Therapy for Critically-Ill COVID-19 Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISMMSCCOVID19
Record Dates: First submitted 2020-05-27; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: COVID; Pulmonary Infection; Sars-CoV2
Keywords: Covid-19 Pneumonia; SARS-CoV-2; Mesenchymal Stem Cells; Umbilical Cord
MeSH Terms: interventions — Oseltamivir; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients receive standardized treatment, consisting of Oseltamivir and Azithromycin
  Interventions: Drug: Oseltamivir; Drug: Azithromycin
- Experiment Group (Experimental): Patients receive intravenous infusion of 1x10^6 unit of umbilical-cord derived mesenchymal stem cells (UC-MSCs)/kgBW in 100 cc of 0.9% NaCl for 1 hour, in addition to standardized treatment
  Interventions: Drug: Oseltamivir; Drug: Azithromycin; Biological: Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Drug: Oseltamivir — Current standardized treatment for Covid-19
Drug: Azithromycin — Current standardized treatment for Covid-19
Biological: Umbilical Cord Mesenchymal Stem Cells — Adjuvant therapy on top of current standardized treatment (Oseltamivir + Azithromycin)
  Arms: Experiment Group

SUMMARY:
Novel Coronavirus (2019nCoV) or Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) that causes Coronavirus Disease 2019, or known as Covid-19 has recently become a global health emergency since it was first detected in Wuhan, the People Republic of China in December 2019. Since then, the prevalence has rapidly increased worldwide. In Indonesia, by the end of April 2020, around 10,000 patients have been tested positive for Covid-19 infection, with a case fatality rate of around 8%.

The pathogenesis of Covid-19 is still under investigation and to our understanding, ACE2 receptors in the alveoli serve as the binding site of the S-protein of envelope spike virus of SARS-CoV-2. TMPRSS2 enzyme aids the fusion between cell membrane and capsid of the virus, allowing penetration of virus into the cell. Vesicles containing virion fuse with cell membrane and released as new virions. Cytopathic effect of the virus and its ability to overcome immune response determines the degree of infection.

Differences in immunological profile among degrees of severity of Covid-19 may vary especially for the number of pro-inflammatory cytokines such as tumor necrosis factor alpha (TNF-α), interleukin (IL)-1, IL-6, IL-8, leukemia-inhibiting factors (LIF), immunological markers such as CXCR3+CD4+, CXCR3+CD8+ T cell and CXCR3+ NK cells, implying the ongoing cytokine storm. The previous studies also found increasing number for infection markers such as procalcitonin, ferritin, and C-reactive protein. The decreasing number of anti-inflammatory cytokines in such as IL-10 also supports this finding.

Previous studies have shown immunomodulating and anti-inflammatory capacity of the mesenchymal stem cells (MSCs). MSCs contributed to the shifting of pro-inflammatory Th2 into anti-inflammatory Th2. One of the most recent study on the usage of MSCs on Covid-19 patients showed increased expression of leukemia inhibitory factor (LIF), which give rise to inhibitory effect of T lymphocyte and natural killer (NK) cell population. Vascular epithelial growth factor (VEGF) is found increasing following MSCs administration, which indicates the ability to improve the disrupted capillaries due to SARS-Cov-2 infection. The ability of MSCs in differentiating to alveolar cells is proven by the presence of SPM and SPC2, surfactant proteins produced by type II alveolar cells. MSCs are unable to be infected by SARS-CoV-2 since they don't have ACE2 receptors and TMPRSS2 enzyme.

DETAILED DESCRIPTION:
This study is a double blind, randomized control trial (RCT). This study will be concluded in 2 months, from May to July 2020, from subject selection to the end of follow up. Research subjects are obtained consecutively from Covid-19 patients who receive care in the intensive care unit (ICU) across four Covid-19 referral hospitals, including Persahabatan Hospital, Sulianti Saroso Center for Infectious Disease, Cipto Mangunkusumo General Hospital, and Universitas Indonesia Hospital, with 10 subjects obtained from each hospital and total 40 subjects for this RCT. Subjects from each hospitals are divided into control and experimental groups. Subject belongs to the control group will receive standardized therapy (consisting of oseltamivir and azithromycin), whereas subjects in the experimental group will receive MSCs infusion, in addition to standardized therapy.

Subject Criteria Inclusion Criteria for MSC Donor from Umbilical Cord:

Umbilical cord is collected from elective caesarean section from a fullterm pregnancies without any complication and free from HIV, Hepatitis B, C, D virus, Cytomegalovirus, Rubella Virus, and free from fungal and bacterial contamination.

Informed consent all of the subjects must be filled and signed up before ruled in this study.

As soon as after delivery, the umbilical cord is collected and processed in sterile specimen 0,9% NaCl at 4oC for 8 hours. The umbilical cord transported to the laboratory and cultured in GMP lab, at Stem Cells Medical Technology Integrated Service Unit Cipto Mangunkusumo Hospital. Cellular viability and proliferation are evaluated after cell characterization test by flow cytometer.

Sterility tests are done three times to ensure cellular sterility. Subjects will receive MSCs through infusion through intravenous for 1 hour, following the administration of diphenhydramine and anticoagulant to prevent clotting.

Following the MSCs administration, monitoring at the patients is carried out every day, whereas laboratory testing for basic parameters (complete blood count, differential count, blood gas analysis, C-reactive protein, SGOT/SGPT (AST/ALT), Ureum/Creatinine, eGFR, electrolyte, procalcitonin, albumin, total bilirubin, D-Dimer, fibrinogen, troponin I and proBNP) are carried out every three days. Cytokine levels are measured before the administration and 7th day after the administration. Chest radiography is carried out every three days.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-95 years old
* Confirmed for diagnosis of Covid-19 through RT-PCR from nasopharyngeal swab and/or bronchoalveolar lavage for patients under intubation
* Laboratory results showed leukopenia and lymphopenic
* Chest radiography shows pneumonia appearance and/or ground-glass opacity on chest CT-Scan
* Patients/their families are willing to sign the informed consent

Exclusion Criteria:

* History of malignancy
* Pregnant, or show positive result on pregnancy test
* Patients was/are currently participating in other clinical trials within the last 3 months

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement: Presence of dyspnea | 15 days
  Assessing whether the patients still have dyspnea, one of cardinal symptoms of Covid-19, assessed from the respiratory rate
Clinical improvement: presence of sputum | 15 days
  Assessing whether the patients still have productive cough, one of cardinal symptoms of Covid-19, assessed from lung auscultation
Clinical improvement: fever | 15 days
  Assessing the presence of fever from measurement of body temperature checking, assessed on daily basis
Clinical improvement: ventilation status | 15 days
  Assessing whether the patients still require ventilation, one of cardinal symptoms of ARDS in Covid-19, assessed from patients' ability during ventilation weaning phase
Clinical improvement: blood pressure | 15 days
  Assessing the patients' blood pressure on daily basis
Clinical improvement: heart rate | 15 days
  Assessing the patients' heart rate on daily basis
Clinical improvement: respiratory rate | 15 days
  Assessing the patients' respiratory rate on daily basis
Clinical improvement: oxygen saturation | 15 days
  Assessing the patients' oxygen saturation on daily basis

SECONDARY OUTCOMES:
General laboratory outcome from leukocyte level | 15 days
  Assessing the changes in total leukocyte upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from lymphocytes level | 15 days
  Assessing the changes in lymphocytes level upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from blood pH | 15 days
  Assessing the changes in blood pH level upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from blood level of CO2 | 15 days
  Assessing the changes in blood pH level upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from blood base excess level | 15 days
  Assessing the changes in blood base excess level upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from blood oxygen partial pressure | 15 days
  Assessing the changes in blood oxygen partial pressure upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from blood level of HCO3 | 15 days
  Assessing the changes in blood level of HCO3 upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from blood level of O2 saturation | 15 days
  Assessing the changes in blood level of O2 saturation upon MSCs administration, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from level of CRP | 15 days
  Assessing the changes in level of CRP, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from level of SGOT/SGPT (AST/ALT) | 15 days
  Assessing the changes in laboratory parameter, consist of SGOT/SGPT (AST/ALT) level, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from the level of ureum/creatinine level | 15 days
  Assessing the changes in laboratory parameter, consist of ureum/creatinine level, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from the level of eGFR | 15 days
  Assessing the changes in laboratory parameter, consist of eGFR, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from the level of sodium | 15 days
  Assessing the changes in level of sodium, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from the level of potassium | 15 days
  Assessing the changes in level of potassium, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from the level of chloride | 15 days
  Assessing the changes in level of chloride, assessed prior to and 1st day after implantation, then once every 3 days post implantation
Changes in procalcitonin level | 15 days
  Assessing the changes in procalcitonin level to assess the anti-inflammatory properties of MSCs, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from albumin level | 15 days
  Assessing the changes in albumin level, assessed prior to and 1st day after implantation, then once every 3 days post implantation
General laboratory outcome from total bilirubin level | 15 days
  Assessing the changes in total bilirubin level, assessed prior to and 1st day after implantation, then once every 3 days post implantation
Changes in D-Dimer level | 15 days
  Assessing the changes in D-Dimer to assess the anti-inflammatory properties of MSCs, assessed prior to and 1st day after implantation, then once every 3 days post implantation
Changes in fibrinogen level | 15 days
  Assessing the changes in fibrinogen to assess the anti-inflammatory properties of MSCs, assessed prior to and 1st day after implantation, then once every 3 days post implantation
Cardiac changes from troponin level | 15 days
  Assessing the changes in troponin level to assess the anti-inflammatory properties of MSCs and their effect in cardiac remodelling, assessed prior to and 1st day after implantation, then once every 3 days post implantation
Cardiac changes from NT proBNP level | 15 days
  Assessing the changes in NT proBNP to assess the anti-inflammatory properties of MSCs and their effect in cardiac remodelling, assessed prior to and 1st day after implantation, then once every 3 days post implantation
Changes in Leukemia Inhibiting Factor | 7 days
  Assessing the changes in leukemia inhibiting factor (LIF) to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of IL-6 | 7 days
  Assessing the changes in level of IL-6 to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of IL-10 | 7 days
  Assessing the changes in level of IL-10 to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of vascular endothelial growth factor (VEGF) | 7 days
  Assessing the changes in vascular endothelial growth factor (VEGF) to assess the effect of growth factors in the MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of ferritin | 7 days
  Assessing the changes in level of ferritin to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of CXCR3 | 7 days
  Assessing the changes in level of CXCR3 to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of CD4 | 7 days
  Assessing the changes in level of CD4 to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of CD8 | 7 days
  Assessing the changes in level of CD8 to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Changes in level of CD56 | 7 days
  Assessing the changes in CD56 to assess the anti-inflammatory properties of MSCs, assessed prior to implantation and on the 7th day post-implantation
Radiologic Improvement from Chest X-Ray/CT Scan | 15 days
  Assessing the changes in radiology examination (Chest X-Ray/CT Scan) for any increased in lung infiltration or ground glass opacity, assessed prior to implantation and once every 3 days post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Ismail H Dilogo, MD, PhD, Principal Investigator — Indonesia University
Locations (4):
- Indonesia (4):
  - Persahabatan General Hospital, Jakarta, DKI Jakarta
  - Sulianti Saroso Center for Infectious Disease, Jakarta, DKI Jakarta
  - Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta
  - Universitas Indonesia Hospital, Depok, West Java